CLINICAL TRIAL: NCT02977585
Title: Helmet Continous Positive Airway Pressure (CPAP) Management and Positive End Expiratory Pressure (PEEP) Level Impact on Severe Bronchiolitis Admitted in Pediatric Intensive Care Units (PICUs)
Brief Title: Helmet Continuous Positive Airway Pressure Support for Severe Bronchiolitis in PICUs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 PANDEMIA
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Emanuele Rossetti, md, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1239_OPBG_2016
Record Dates: First submitted 2016-11-17; First posted 2016-11-30 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Critically Ill Severe Bronchiolitis
Keywords: continous positive airway pressure; helmet; non invasive; positive end expiratory pressure; severe bronchiolitis; pediatric intensive care unit
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): high level support
  Interventions: Device: 10 cmH2O peep
- group 0 (No Intervention): low level support

INTERVENTIONS:
Device: 10 cmH2O peep — positive end expiratory pressure
  Arms: group 1

SUMMARY:
Binary randomized peep level of Helmet CPAP (1-0). The first patient enrolled will be assign to treatment 1 (10 cmH2O peep level), independently from its BSS. The following patients enrolled will be assign to treatment 0 (5 cmH2O peep level), and consecutively up to 25 patients at least.

* 10 cmH2O peep, 50 L/min gas flow, fraction of inspired oxygen (FiO2) 0.5 on PICU admission (random 1)
* 5 cmH2O peep, 50 L/min gas flow, FiO2 0.5 on PICU admission (random 0) If clinical and respiratory worsening, reduction of pH or partial oxygen arterial pressure (PaO2)/FiO2 occurs in the following first hour after Helmet CPAP treatment start, patients enrolled will receive endotracheal intubation, full face mask non invasive ventilation or higher peep level treatment (7.5-10 cmH2O) according to clinical evaluation, if necessary.

In investigator's experience, early worsening of severe bronchiolitis in PICU in the first hour of Helmet CPAP treatment with 10 cmH2O peep level leads to endotracheal intubation.

DETAILED DESCRIPTION:
INTRODUCTION

Newborns and infants with severe bronchiolitis admitted in PICU (Pediatric Intensive Care Unit) are patients at high risk for invasive mechanical ventilation support. In current literature, there is lack of multicenter, prospective and randomized studies to assess and describe the impact of non invasive ventilation support among severe bronchiolitis admitted in PICU, notwithstanding the actual improvement of non invasive ventilation technique on intubation rate reduction.

Recently, we can find studies on bronchiolitis management in pediatric ward and supported with high flow nasal cannula (HFNC).

The studies on severe bronchiolitis admitted in PICU do not evaluate positive end expiratory pressure (Peep) level applied during Helmet continous positive airway pressure (CPAP) support.

According to Italian PICU Network (TIPNET) data, severe bronchiolitis admitted in PICU intubation rate is close to 10% (report 2010-2016), whatever non invasive ventilation support has been used.

Principal investigators have performed a retrospective and cohort chart review among severe bronchiolitis (82) admitted in PICU from 2011 to 2015. Early Helmet CPAP was applied to patients, but peep level has been provided according to clinician experience, because of lack of indication on this issue. Patients were admitted in PICU from Emergency department, pediatric ward and up to 72 hours of ineffective HFNC support. The investigators have studied intubation rate, length of stay, bronchiolitis severity score, virus infection, peep level and gas flow applied on Helmet CPAP.

According to preliminary results, 10 cmH2O peep level results 50 time more protective than lower (5-7.5 cmH2O) peep among flow rate of 50 L/min.

Intubation rate with peep level 10 cmH2O was 3%, while it rose over 15% among 7.5-5 cmH2O peep level. Statistically significant difference were found on length of PICU stay.

Scientific literature on Helmet CPAP noising exposure is poor. Such noising was proved to be reduced with filter application on Helmet CPAP respiratory circuit. There are not report, and we have never experienced acoustic system impairment in patients undergone Helmet CPAP.

AIMS Primary aim: to evaluate escalation therapy (higher peep, non invasive ventilation in pressure support mode, or intubation and mechanical ventilation) rate on severe bronchiolitis admitted in PICU and supported with Helmet CPAP non invasive ventilation with 10 cmH2O peep level in group 1, and 5 cmH2O peep level in group 0.

Secondary aim: to evaluate, among two study groups, length of PICU stay, pneumothorax incidence on Helmet CPAP, sedation effect during Helmet CPAP, early enteral feeding tolerance, syncytial and other respiratory virus incidence, bacterial infection and 30 days outcome.

DESIGN Prospective, randomized, cohort, controlled and multicentric study.

Population: sample size The study requires 488 patients, enrolled among 20 national and international PICU. Sample size have been calculated on preliminary results of our retrospective chart review; we hypothesize that intubation rate with 5 cmH2O peep level is 15% and application of 10 cmH2O peep level may reduce it to 50%. According to these hypothesis, we need 244 patients for each group to have 5% of significativity level and 80% of study power.

Length of study 24 months

Procedure and methods

Selection and patient enrollment Severe bronchiolitis admitted in PICU and requiring respiratory support.

Intervention

Binary randomized peep level of Helmet CPAP (1-0). The first patient enrolled will be assign to treatment 1 (10 cmH2O peep level), independently from its BSS. The following patients enrolled will be assign to treatment 0 (5 cmH2O peep level), and consecutively up to 25 patients at least.

* 10 cmH2O peep, 50 L/min gas flow, FiO2 0.5 on PICU admission (random 1)
* 5 cmH2O peep, 50 L/min gas flow, FiO2 0.5 on PICU admission (random 0) If clinical and respiratory worsening, reduction of pH or PaO2/FiO2 occurs in the following first hour after Helmet CPAP treatment start, patients enrolled will receive endotracheal intubation, full face mask non invasive ventilation or higher peep level treatment (7.5-10 cmH2O) according to clinical evaluation, if necessary.

In investigators' experience, early worsening of severe bronchiolitis in PICU in the first hour of Helmet CPAP treatment with 10 cmH2O peep level leads to endotracheal intubation.

STUDY PLAN Application of a standard treatment protocol for all patients enrolled. It is the same standard of care applied to treat these patients in our PICU in the last 2 years. Of course, patients who will not be enrolled in the study will be supported and treated with the best feasible care.

* Registration of the modified Wood's Clinical Asthma score (mWCAS) for severe bronchiolitis admitted in PICU (Bronchiolitis Severity Score-BSS)
* clarithromycin prophylaxis for newborns (up to 30 days old), or I generation cephalosporine for older infants, if high fever, lung opacities or high inflammation markers occurs (PCR, procalcitonin, White body cells)
* volume replacement (20 ml/kg of sodium chloride solution or albumine 5%) in 60 min
* morphine ev bolus: 20 mcg/kg in 2 min and following 5 mcg/kg/h infusion (or other sedatives according to local PICU investigator)
* nasogastric tube placement and early enteral feeding 4-6 hours after admission (5-10 ml/h)
* desamethasone 0.2 mg/kg x3/die ev (according to local PICU investigator ).
* proton pump inhibitors or H2 receptor antagonist (according to local PICU investigator).
* aerosol therapy 4 time/die: sodium chloride hypertonic solution 3% (or sodium chloride 0.9%) 2 ml with ipratropium bromide .
* Arterial blood gas exam (ABE) before Helmet CPAP application and in the following 1,12 24, and 48 hours; arterial catheter positioning is preferred (or arterial blood sampling by direct arterial puncture according to local PICU practice).
* Pharyngeal swab for molecular analysis to detect viral DNA will be performed on PICU admission, if not yet performed.
* occipital and neck skin protection will be used to avoid Helmet CPAP pressure sores.
* each Helmet will be provided of a filter to reduce noise inside it.
* Helmet gas will flow through heat-moisture device switched on 5 min/hour

Only patients whose parents have signed written informed consent will be enrolled in this study. Any direct follow up is supposed after PICU discharge. Monitoring of hospital discharge will be followed by intranet database of the participant hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 38 weeks of gestational age up to 18 months old, admitted in PICU for severe bronchiolitis, whose parents have signed written informed consent to enroll the child in the study.
* Patients with severe bronchiolitis moved from emergency department, pediatric ward, and supported up to 72 hours with HFNC or O2 therapy.

Exclusion Criteria:

* Severe congenital malformation Inborn congenital error Neonatal or postnatal neurologic disorder Parents refusal to study participation Presence or supposed pneumothorax on chest X-ray or lung ultrasound

Ages: 38 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
incidence of intubation following Helmet CPAP treatment | 7 days
  to evaluate intubation rate on severe bronchiolitis admitted in PICU and supported with Helmet CPAP non invasive ventilation with 10 peep level in group 1, and 5 peep level in group 0.
incidence of pneumothorax following Helmet CPAP treatment | 72 hours
  pneumothorax occurrence

SECONDARY OUTCOMES:
length of stay | days 30
  length of PICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Children's Hospital, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Donlan M, Fontela PS, Puligandla PS. Use of continuous positive airway pressure (CPAP) in acute viral bronchiolitis: a systematic review. Pediatr Pulmonol. 2011 Aug;46(8):736-46. doi: 10.1002/ppul.21483. Epub 2011 May 26. PMID 21618716
- [Background] Mayfield S, Bogossian F, O'Malley L, Schibler A. High-flow nasal cannula oxygen therapy for infants with bronchiolitis: pilot study. J Paediatr Child Health. 2014 May;50(5):373-8. doi: 10.1111/jpc.12509. Epub 2014 Feb 25. PMID 24612137
- [Background] Trevisanuto D, Camiletti L, Doglioni N, Cavallin F, Udilano A, Zanardo V. Noise exposure is increased with neonatal helmet CPAP in comparison with conventional nasal CPAP. Acta Anaesthesiol Scand. 2011 Jan;55(1):35-8. doi: 10.1111/j.1399-6576.2010.02356.x. Epub 2010 Nov 15. PMID 21077846
- [Background] Chidini G, Piastra M, Marchesi T, De Luca D, Napolitano L, Salvo I, Wolfler A, Pelosi P, Damasco M, Conti G, Calderini E. Continuous positive airway pressure with helmet versus mask in infants with bronchiolitis: an RCT. Pediatrics. 2015 Apr;135(4):e868-75. doi: 10.1542/peds.2014-1142. Epub 2015 Mar 16. PMID 25780074
- [Background] Ganu SS, Gautam A, Wilkins B, Egan J. Increase in use of non-invasive ventilation for infants with severe bronchiolitis is associated with decline in intubation rates over a decade. Intensive Care Med. 2012 Jul;38(7):1177-83. doi: 10.1007/s00134-012-2566-4. Epub 2012 Apr 18. PMID 22527081
- [Background] Milani GP, Plebani AM, Arturi E, Brusa D, Esposito S, Dell'Era L, Laicini EA, Consonni D, Agostoni C, Fossali EF. Using a high-flow nasal cannula provided superior results to low-flow oxygen delivery in moderate to severe bronchiolitis. Acta Paediatr. 2016 Aug;105(8):e368-72. doi: 10.1111/apa.13444. Epub 2016 May 16. PMID 27102726
- [Background] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575